CLINICAL TRIAL: NCT02831335
Title: Technical Development of Multi-Parametric Renocerebral MRI
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1603M85492
Record Dates: First submitted 2016-06-15; First posted 2016-07-13 (Estimated); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Group 1: normal 21-35 years old participants
  Interventions: Other: MRI
- Group 2: normal 36-50 years old participants
  Interventions: Other: MRI
- Group 3: normal 51-65 years old participants
  Interventions: Other: MRI
- Group 4: normal 66- 80 years old participants
  Interventions: Other: Group 4

INTERVENTIONS:
Other: MRI — Perform MRI studies
  Groups: Group 1
Other: MRI — Perform MRI studies
  Groups: Group 2
Other: MRI — Perform MRI studies
  Groups: Group 3
Other: Group 4 — Perform MRI studies
  Groups: Group 4

SUMMARY:
The purpose of the study is to investigate the associations of the age-related changes in the brain, kidneys and cognitive performance in healthy adults by utilizing multiple anatomic and functional MRI methods along with a battery of cognitive tests.

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking as primary language
2. No hearing loss or uncorrected vision

Exclusion Criteria:

1. Lacking capacity to consent
2. Having known history of cardiovascular diseases (e.g., clinical stroke)
3. Having acute and chronic obstructive pulmonary disease
4. Having known history of renal diseases (e.g., acute kidney injury)
5. Having known history of cognitive disorder or psychiatric illness
6. Having known history of chemical dependence (e.g., alcohol and narcotics)
7. Being treated with stimulant medications, anticonvulsants, antihypertensives or ß-adrenergic blockers

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal participants will be recruited for four age groups with the following age ranges: 21 - 35, 36 -50, 51 - 65 and 66 - 80 years. For each subject group, equal number of male and female subjects will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
MRI measured perfusion for each group | Baseline
  MRI measurements will be summarized for each group by using mean and standard deviation or standard error.
MRI measured vascular reactivity for each group | Baseline
  MRI measurements will be summarized for each group by using mean and standard deviation or standard error.
Cognitive performance for each group | Baseline
  The total cognitive performance scores will be summarized for each group by using mean and standard deviation or standard error.

CONTACTS AND LOCATIONS:
Overall Officials: Xiufeng Li, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- Center for Magnetic Resonance Research, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No